CLINICAL TRIAL: NCT05907681
Title: Prospective Observational Study on Outcome of High-precision Hypo-fractionated Radiotherapy in Metastatic Breast Cancer (PRECISE-M)
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Haeyoung Kim, Associate professor, Samsung Medical Center
Other Study IDs: 2023-04-032-003
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Radiation Therapy Complication
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective observational study on outcomes of high precision hypo-fractionated radiotherapy in breast cancer with distant metastasis.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed breast cancer
* presence of distant metastasis
* radiation therapy using IMRT, SBRT, or proton therapy is done or planned
* Able and willing to comply with the study protocol

Exclusion Criteria:

* unable to adhere to the study protocol

Ages: 19 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women treated with hypofractionated RT using IMRT, SBRT, or proton therapy for metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Local control rate | 1-year
  LC after radiation therapy

SECONDARY OUTCOMES:
Overall survival rate | 1-year
Disease-free survival | 1-year
  disease-free survival rate after the time of RT
Treatment-related toxicities | 1-year
  Acute and chronic radiation toxicities according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Haeyoung Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided